CLINICAL TRIAL: NCT06902155
Title: Impact of Diabetes Subtypes on Urinary Incontinence During Pregnancy and Postpartum: A Study on BMI and Glycemic Control
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Cam ve Sakura Sehir Hastanesi
Record Dates: First submitted 2025-03-21; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Urinary Incontinence; Diabetes Mellitus
Keywords: Urinary incontinence; pregnancy; diabetes mellitus; Body mass index; glycemic control.
MeSH Terms: conditions — Urinary Incontinence; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- T1DM group: type 1 diabetes mellitus group (n = 16)
  Interventions: Diagnostic Test: International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF)
- T2DM group: type 2 diabetes mellitus group (n = 32)
  Interventions: Diagnostic Test: International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF)
- GDM group: gestational diabetes mellitus group (n = 51)
  Interventions: Diagnostic Test: International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF)
- control group (CG): consisting of healthy pregnant women with uncomplicated pregnancies (n = 48).
  Interventions: Diagnostic Test: International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF)

INTERVENTIONS:
Diagnostic Test: International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) — Urinary incontinence was assessed using the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), a validated instrument with a Cronbach's alpha of 0.88. This tool consists of four items: three scored questions evaluating leakage frequency (0-5), volume (0-6), and impact on quality of life (0-10), summing to a total score of 0-21, and one unscored question identifying situations where incontinence occurs. Two separate analyses were performed: total ICIQ-SF score and responses to question, which identified UI-triggering situations

SUMMARY:
Objective: This study investigated the relationship between diabetes mellitus and urinary incontinence (UI) during pregnancy and postpartum, focusing on metabolic factors like body mass index (BMI) and glycemic control.

Methods: A prospective observational study was conducted at Başakşehir Çam and Sakura City Hospital, including 147 pregnant women in their third trimester (≥30 weeks). Participants were categorized into type 1 diabetes mellitus (n = 16), type 2 diabetes mellitus (n = 32), gestational diabetes mellitus (GDM) (n = 51), and a control group (n = 48). UI was assessed using the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), and metabolic parameters were retrieved from hospital records. Subgroup comparisons and ROC curve analysis were performed to determine BMI and HbA1c cut-off values for predicting postpartum UI.

DETAILED DESCRIPTION:
This prospective observational study was conducted at …… between ……with participants recruited from the obstetrics department. A total of 147 pregnant women in their third trimester (≥30 weeks) were enrolled and categorized into four groups: type 1 diabetes mellitus (T1DM) group (n = 16), type 2 diabetes mellitus (T2DM) group (n = 32), gestational diabetes mellitus (GDM) group (n = 51), and a control group (CG) consisting of healthy pregnant women with uncomplicated pregnancies (n = 48). Participants were aged between 18 and 40 years and had good physical and mental health. Eligibility criteria included singleton pregnancy, gestational age of at least 30 weeks, and no history of known urological disorders, while exclusion criteria encompassed multiple pregnancies, chronic kidney disease, and prior urogynecological surgery.

Maternal age, insulin use, and history of pre-pregnancy urinary incontinence (UI) were obtained through direct patient interviews. Third-trimester HbA1c levels and complete urinalysis results were extracted from the hospital's digital medical records. Urinary incontinence was assessed using the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), a validated instrument with a Cronbach's alpha of 0.88. This tool consists of four items: three scored questions evaluating leakage frequency (0-5), volume (0-6), and impact on quality of life (0-10), summing to a total score of 0-21, and one unscored question identifying situations where incontinence occurs. Two separate analyses were performed: total ICIQ-SF score and responses to question 6, which identified UI-triggering situations.

To minimize selection bias, only participants meeting strict inclusion and exclusion criteria were enrolled. The study size was determined based on previous studies to ensure adequate statistical power for subgroup analyses.

ELIGIBILITY:
Inclusion Criteria:).

1. Aged between 18 and 40 years
2. Had good physical and mental health.
3. Had singleton pregnancy
4. Had no history of known urological disorders
5. At least 30 weeks gestational aged , pregnants

Exclusion Criteria:

1. multiple pregnancies
2. pregnants with chronic kidney disease, and prior urogynecological surgery.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: This study included a total of 147 pregnant women in their third trimester (≥30 weeks) recruited from the obstetrics department. Participants were categorized into four groups: type 1 diabetes mellitus (T1DM) (n = 16), type 2 diabetes mellitus (T2DM) (n = 32), gestational diabetes mellitus (GDM) (n = 51), and a control group (CG) comprising healthy pregnant women with uncomplicated pregnancies (n = 48). Eligible participants were aged between 18 and 40 years and in good physical and mental health. Inclusion criteria required a singleton pregnancy with a gestational age of at least 30 weeks and no history of known urological disorders. Exclusion criteria included multiple pregnancies, chronic kidney disease, and prior urogynecological surgery.
Sampling Method: Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Maternal serum HbA1c levels for pregnancy-related and postpartum UI | From the time of inclusion in the study until the first postpartum month.
  HbA1c levels were significantly associated with an increased severity of incontinence in women with GDM.
BMI for pregnancy-related and postpartum UI | From the time of inclusion in the study until the first postpartum month.
  BMI was a strong predictor of postpartum incontinence persistence in both the type 1 diabetes and GDM groups,
insulin use for pregnancy-related and postpartum UI | From the time of inclusion in the study until the first postpartum month.
  insulin use did not significantly impact UI severity during pregnancy in any of the diabetes subgroups.
maternal age and history of urinary tract infection for pregnancy-related and postpartum UI | From the time of inclusion in the study until the first postpartum month.
  maternal age and history of urinary tract infection were not significantly associated with UI severity or postpartum incontinence in any diabetes group.

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam ve Sakura Sehir Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vesentini G, Piculo F, Marini G, Barbosa AMP, Corrente JE, Rudge MVC. Impact of Obesity and Hyperglycemia on Pregnancy-specific Urinary Incontinence. Rev Bras Ginecol Obstet. 2023 Jun;45(6):303-311. doi: 10.1055/s-0043-1770087. Epub 2023 Jul 21. PMID 37494572
- [Result] Valerio PM, Zordao CC, Goncalves VE, Hasegawa MSR, Jorge CH, Moises ECD, de Oliveira Guirro EC. Urinary Incontinence in the Third Trimester of Pregnancy of Type 1 Diabetic Women. Reprod Sci. 2024 Jun;31(6):1558-1564. doi: 10.1007/s43032-024-01488-w. Epub 2024 Mar 4. PMID 38438778